CLINICAL TRIAL: NCT02831868
Title: Multi Center, Open-label, Single Arm, Study Designed to Evaluate Safety, Tolerability and Efficacy of HAVAI, a Minimally Invasive Implant Composed of Spring, Double Anchor and Suture, Versus Standard of Care 1st Metatarsal Osteotomy, for Correction of Inter-metatarsal Angle in Subjects Suffering From Hallux Valgus Deformity
Brief Title: Safety, Tolerability and Efficacy of HAVAI, for Correction of Inter-metatarsal Angle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 415-16
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-03

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXP (Experimental): Implantation of a HAVAI device to correct HVA without osteotomy
  Interventions: Device: HAVAI

INTERVENTIONS:
Device: HAVAI — implantation of the HAVAI device to correct the IMA angle

SUMMARY:
A non-inferiority study to demonstrate efficacy of the HAVAI minimally invasive device compared to standard of surgical care 1st metatarsal osteotomy (SSOC)

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and female subjects, aged 20 to 75 years old, inclusive, at screening visit.
2. Subject weighing <100 kg and body mass index (BMI) <32 kg/m2.
3. Subjects with confirmed diagnosis of HV deformity based on radiography assessment of IMA 12°-15°.
4. Able and willing to comply with the requirements of the protocol.
5. Able to understand and sign written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who need or may need to have 2nd MT osteotomy as part of their index surgery (e.g. instability or subluxation of 2nd MTPJ)
2. History of:

   a. Severe Diabetes mellitus (defined as existence of: i. More than 10 years duration ii. HbA1C 8.0 < iii. any known complications of diabetes (PVD, Nephropathy [CR>1.3], retinopathy, IHD)) b. Claudication, known peripheral vascular disease or no palpable pulses (DP or TP).

   c. Known rheumatoid or inflammatory disease. d. X-ray evidence of moderate osteoarthritis of MTPJ-1 or TMTJ-1. e. neurological conditions associated with spasticity or lower limb paralysis. f. Prior operation on MT1 or MT2. g. Fracture (past or present) of MT1 or MT2.
3. Aseptic necrosis or any deformity of MT2 head.
4. Aseptic necrosis of the MT1 head
5. Pregnant women or women with childbearing potential who are not obliged to take any contraception measures
6. Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agent(s)
7. ASA grade above 2

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
A change in IMA angle | 50 weeks
  A change in IMA angle - compared to baseline using t test for repeated measures with 0.05 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Heller, MD, Principal Investigator — Rabin MC
Locations (2):
- Israel (2):
  - Rambam Hospital, Haifa
  - Bonfix Ltd, Jerusalem

IPD SHARING:
Plan to Share IPD: No